CLINICAL TRIAL: NCT04857242
Title: Electrical Impedance Tomography Measurements During Apnea Test in Patients With Suspected Brain Death
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kiskunhalas Semmelweis Hospital the Teaching Hospital of the University of Szeged (Other Government)
Collaborators: Budapest University of Technology and Economics (Other); Hochschule Furtwangen University (Other); Szeged University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: apnEIT
Record Dates: First submitted 2021-04-22; First posted 2021-04-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Brain Death
Keywords: Apnea testing; Electrical Impedance Tomography
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apnea test, recruitment manoeuvre (Experimental): 1. Continuous electric impedance tomography (EIT) recording. Recording of initial vital parameters and arterial blood gas results. Adjusment of PaCO2 between 38-42 mmHg, 10 minutes of preoxygenation with FiO2 of 1.0 then disconnection of the patient from the ventilator.
  2. Continuous administration of 6 L/min O2 flow via a catheter into the tracheal tube.
  3. Arterial blood gas sampling and recording of vital parameters in every second minutes. Detection of any spontaneous respiratory movement by the apnoe test investigator or by EIT signals.
  4. Reconnection with respirator if there is any sign of spontaneous breathing effort or if there is no spontaneous breathing effort and the PaCO2 is over 60 mmHg. Recording of vital parameters.
  5. Recruitment manoeuvre (PEEP 20 cmH2O, pressure control 20 cmH20 for 40 minutes) then set up of the initial ventilator parameters.
  6. Terminal arterial blood gas results and vital parameters 5 minutes following the end of the recruitment manoeuvre.
  Interventions: Diagnostic Test: Apnea test, alveolar recruitment

INTERVENTIONS:
Diagnostic Test: Apnea test, alveolar recruitment — Alveolar recruitment following the phase of apnea testing

SUMMARY:
Apnea testing is the final decisive examination in the strictly regulated process of brain death assessment. There is no standardized method found in the literature for apnea testing except for the inspection of possible spontaneous chest movements. In addition, the test itself lasts for several minutes leading to the collapse of the lungs.

Electrical impedance tomography (EIT) is a non-invasive, real-time monitoring technique, which is suitable for detecting changes in lung volumes during ventilation. With its help, one can examine the spontaneous initiation of inspiration, the development of atelectasis and the reopening of collapsed regions by mechanical ventilation.

Furthermore, the apnea test provides for analysing the effect of changes in pulmonary perfusion on impedance in the absence of noise generated by ventilation.

DETAILED DESCRIPTION:
The aim of the study is to assess the eligibility of electrical impedance monitoring for the detection of possible spontaneous initiations of inspiration during apnea test in patients with suspected brain death. The study could contribute to the opening of new areas in the clinical use of the electrical impedance device. An additional aim is to observe the collapse and the reopening by recruitment manoeuvers of different pulmonary regions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected brain death undergoing apnea test for detecting the absence of spontaneous breathing

Exclusion Criteria:

* age under 18
* pregnancy
* pulmonectomy, lung resection in the past medical history
* clinically end stage chronic obstructive pulmonary disease (COPD)
* severe hemodynamic instability (vasopressor refractory shock)
* severe bullous emphysema and/or spontaneous pneumothorax in the past medical history
* chest drainage in situ due to pneumothorax and/or bronchopleural fistula

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
detection of spontaneous inspiration | 20 minutes
  Detection of absolute changes in impedance using EIT during apnea test, which may refer to spontaneous initiations of inspiration

SECONDARY OUTCOMES:
Gas exchange | 20 minutes
  Change in arterial partial pressure of oxygen (PaO2) (mmHg) following alveolar recruitment performed after apnea testing
Dynamic compliance | 20 minutes
  Change in dynamic compliance (ml/cmH2O) following alveolar recruitment
End expiratory lung impedance | 20 minutes
  Change in end expiratory lung impedance (EELI) (%) following alveolar recruitment
Center of ventilation | 20 minutes
  Change in center of ventilation (%) following alveolar recruitment
Lung perfusion | 20 minutes
  Changes in lung perfusion during the apnea phase (%)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No